CLINICAL TRIAL: NCT05619471
Title: VIO Imaging for Skin Tissue Assessment (VISTA) - a Prospective, Multicenter Investigation of the VIO Device in Subjects Undergoing Routine Biopsy
Brief Title: VIO Imaging for Skin Tissue Assessment (VISTA)
Acronym: VISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enspectra Health (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR-30096; 2R44CA221591-03 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-11-17 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Skin Condition; Skin Diseases; Skin Lesion; Skin Abnormalities; Skin Cancer
MeSH Terms: conditions — Skin Diseases; Skin Abnormalities; Skin Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- VIO Imaging (Experimental): Subjects with skin conditions that are candidates for biopsy
  Interventions: Device: VIO Imaging

INTERVENTIONS:
Device: VIO Imaging — Skin conditions that are candidates for skin biopsies

SUMMARY:
To demonstrate the safety and effectiveness of the VIO device in obtaining in vivo images that show tissue features including epidermis, dermis, collagen, blood vessels, and/or pigment.

To demonstrate that the tissue features identified on the images obtained with the VIO device align with the corresponding pathology images procured from the skin biopsy.

To evaluate the ability of blinded readers to correctly identify tissue features on images obtained with the VIO device.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is between 18 and 99 years of age.
2. The subject or Legally Authorized Representative (LAR) is able and willing to provide written informed consent.
3. The subject is planning to undergo a routine skin biopsy.
4. The subject is willing and able to remain still for periods of up to 3 minutes to allow for image capture.
5. The subject or LAR has sufficient mental capacity to understand the informed consent form (ICF) and comply with the protocol requirements.

Exclusion Criteria:

1. The subject has a general health condition or systemic disease that in the opinion of the physician, precludes them from trial participation.
2. The subject has a known allergy or increased skin sensitivity to silicone, adhesives, or glycerin.
3. The subject's lesion targeted for biopsy:

   1. Is located on the palms of the hands, soles of the feet, fingernails, or toenails.
   2. Has dense hair that will not be removed prior to the skin biopsy.
   3. Has clinically significant abraded or ulcerated skin with or without discharge.
   4. Is associated with a wound or skin condition that in the opinion of the physician precludes them from participation
   5. Is located in mucosal tissue (i.e., oral, nasal, etc.).
   6. Is on tattooed skin.
   7. Is on a skin formation too tortuous for the investigational device to access (e.g., skin tags.)
   8. Is located in the periorbital region or directly on the eyelid.

      -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wang, MD, FAAD, Principal Investigator — Golden State Dermatology
Locations (2):
- United States (2):
  - Golden State Dermatology, Merced, California
  - Golden State Dermatology, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ward WH, Farma JM, editors. Cutaneous Melanoma: Etiology and Therapy [Internet]. Brisbane (AU): Codon Publications; 2017 Dec 21. Available from http://www.ncbi.nlm.nih.gov/books/NBK481860/ PMID 29461771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period:
  22-Oct-2022 t0 29-Dec-2022
Units Other Than Participants: 65 lesions
Period: Overall Study
Arm/Group | VIO Imaging
Started | 65; 65 65 lesions
Completed | 65; 65 65 lesions
Not Completed | 0; 0 65 lesions

BASELINE CHARACTERISTICS:
Population: Subjects that are planning to undergo a routine skin biopsy
Groups:
- VIO Imaging: Adult subjects between 18 and 99 years of age willing and able to provide written informed consent either themselves or by their legally authorized representative (LAR) and planning to undergo a routine skin biopsy and adhere to study specific requirements.
Arm/Group | VIO Imaging
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a demographic measure of skin pigment and sensitivity to sunlight, as self-reported by participants prior to the study procedure. The measure ranges from Type I (least pigment/most sensitive) to Type VI (most pigment/least sensitive). Refer to PubMed ID: 29461771 for the scale used.
  Participants
    Type I | 6
    Type II | 18
    Type III | 27
    Type IV | 11
    Type V | 3
    Type VI | 0
Anatomical Location [Count of Participants; unit: Participants]
  Head and Neck | 38
  Torso | 6
  Limbs | 21

OUTCOME MEASURES:

1. Primary Outcome: Comparative Reader Percentage Agreement
Description: This outcome measured the % agreement and validation of specific tissue features on VIO images in comparison to gold standard pathology images between N=3 Comparative Readers (CRs). "CRs" were study investigators that were selected based on their experience and medical qualifications. 100% agreement and validation between the CRs was required to proceed to the next study phase.
Time Frame: 8 months post-enrollment completion
Population: Comparative Reader Agreement and Validation was conducted on images taken of all participants
Measure: Number; unit: percentage of agreement
Units Other Than Participants: Images
Groups:
- Training Set: 141 images from 26 subjects (1 lesion per subject) were selected as Training Set Data to evaluate this primary outcome measure
- Validation Set: 248 lesions from 39 subjects (1 lesion per subject) were selected as Validation Set Data to evaluate this primary outcome measure
Arm/Group | Training Set | Validation Set
Number analyzed (Participants) | 26 | 39
Number analyzed (Images) | 141 | 248
percentage of agreement | 100 | 100

2. Primary Outcome: Blinded Reader Percentage Agreement
Description: This outcome measured the % agreement between N=3 Blinded Readers (BRs) of their assessment of VIO images in comparison to the answer key developed from the Comparative Reader validation. "BRs" were study investigators that were selected based on their experience and medical qualifications. >90% agreement was required to proceed to the next study phase.
Time Frame: 8 months post-enrollment completion
Measure: Number; unit: percentage of agreement
Units Other Than Participants: Questions
Groups:
- Performance Test: 450 performance test questions from the Validation Data Set (39 subjects) were generated to evaluate this outcome measure
Arm/Group | Performance Test
Number analyzed (Participants) | 39
Number analyzed (Questions) | 450
percentage of agreement | 94

3. Primary Outcome: Safety / Adverse Events
Description: Safety will be assessed as the incidence of all adverse events (analyzed by severity, seriousness, and relationship to the device and procedure) that occur through the 7-day follow-up period.
Time Frame: 7 +/- 3 days after VIO imaging
Measure: Number; unit: adverse events
Groups:
- All Subjects: All 65 subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 65
adverse events | 0

4. Secondary Outcome: Inter-Reader Percentage Agreement
Description: This outcome measured the inter-reader % agreement between N=3 Blinded Readers (BRs) during image analysis. Minimum 90% agreement was required to proceed to the next study phase.
Time Frame: 8 months post-enrollment completion
Measure: Number; unit: percentage of agreement
Units Other Than Participants: Questions
Arm/Group | Performance Test
Number analyzed (Participants) | 39
Number analyzed (Questions) | 450
percentage of agreement
  Region | 94
  Feature | 93

5. Secondary Outcome: Evaluation of Secondary Histopathology Characteristics
Description: This outcome measured the % agreement between N=3 Blinded Readers (BRs) of their assessment of secondary histopathology characteristics in VIO images in comparison to the answer key developed from the Comparative Reader validation. >90% agreement was required to proceed to the next study phase.
Time Frame: 8 months post-enrollment completion
Population: Performance testing on secondary features (Stratum corneum, Hair shaft or follicle, Solar elastosis, Hyperkeratosis, Nodule or nest of cells, Atypia, Epidermal disarray) was conducted using 179 test questions
Measure: Number; unit: percentage of agreement
Units Other Than Participants: Questions
Groups:
- Performance Test (Secondary Features): 179 performance test questions for secondary features (out of 450 total) from the Validation Data Set (39 subjects) were generated to evaluate this outcome measure
Arm/Group | Performance Test (Secondary Features)
Number analyzed (Participants) | 39
Number analyzed (Questions) | 179
percentage of agreement | 98

ADVERSE EVENTS:
Time Frame: 7+/-3 days after enrollment
Description: See clinicaltrials.gov definition
Groups:
- VIO Imaging: Adult subjects with skin conditions that are candidates for routine skin biopsies
Arm/Group | VIO Imaging
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consultant (PI) shall not, either during or subsequent to the Term of the Agreement, directly or indirectly publish any such information (Proprietary Information) without the prior written authorization from Company (Sponsor).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT05619471/Prot_SAP_000.pdf